CLINICAL TRIAL: NCT06722144
Title: Animal-assisted Therapy Improves Cognitive and Emotion in Nursing Home Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-02-014C
Record Dates: First submitted 2024-04-30; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Supportive Care; Treatment; Prevention
Keywords: behavioral and psychological symptoms; animal assisted therapy; cognition
MeSH Terms: conditions — Behavior | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Nursing home residents were dementia and older.
Who Masked: Participant
Masking Description: There are blinding of participants and their family.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- emotion status (Experimental): Geriatric Depression Scale and Short Form Health Scale(GDS-15)
  Interventions: Behavioral: Animal-assisted Therapy
- cognition status (Experimental): Short Portable mental state questionnaire(SPMSQ)
  Interventions: Behavioral: Animal-assisted Therapy
- feeling healthy (Experimental): Brief Symptom Rating Scale(BSRS-5)
  Interventions: Behavioral: Animal-assisted Therapy
- activities of daily living status (Experimental): Barthel index scale
  Interventions: Behavioral: Animal-assisted Therapy

INTERVENTIONS:
Behavioral: Animal-assisted Therapy — By the professor leader makes social interaction, and helping residents with rehabilitation through the Doctor dogs.
  Other Names: pet therapy; the doctor dog

SUMMARY:
More than 80% of the residents of the investigator's nursing home are dementia, who are often mentally and emotionally unstable. The staff need to spend time helping to eliminate problems. The investigator assume that non-drug intervention measures can be added, such as the Animal-assisted Therapy (AAT). The hypothesis for ATT is expected to improve the mental and emotional inappropriate manifestations of dementia, reduce interfering behaviors, improve the quality of life, reduce the use of inappropriate mental drugs, and expect residents to delay the degradation of physiological functions.

DETAILED DESCRIPTION:
Nursing homes in the investigator's country accept dementia residents usually. The dementia residents often suffer from mental and emotional problems. Then they used drugs to improve the mental and emotional conditions. There were many studies about non-drug treatments ,such as: gardening, nostalgia, pets, and other interventions were improved for the mental and emotional to dementia residents.Well-trained therapy dogs exhibit the behavior that human patients construe as friendly and welcoming.AAT dogs are also required to possess a calm temperament for accommodating the contact with unfamiliar clients while they serve as a source of comfort. In domestic observational studies, non-pharmaceutical interventions for people with dementia who have activities and the hypothesis for ATT can improve the quality of care for dementia, reduce the use of mentally inappropriate drugs, and delay the degree of degeneration. Recent evidence has shown that nursing institutions with dementia arranged weekly activities with AAT for a period of 6 months. Significant improvement was in social interaction, emotional expression, and behavioral and psychological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Residents of long-term care homes
* No fear or allergy to dogs
* Wheelchair accessible persons
* Able to communicate in Mandarin and Taiwanese
* Agree to sign the subject consent form

Exclusion Criteria:

* Non-residents of nursing homes
* Fear and allergy to dogs
* Bedridden and wheelchair users
* Do not agree to sign the subject consent form

Note: Although many nursing home residents have symptoms of dementia, many have not been diagnosed by a doctor, so dementia and other related diseases cannot be included in the inclusion or exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
The Short Portable mental state questionnaire (SPMSQ) | The experimental and control groups were subjected to a pre-test after they were recruited. There are 12 times AAT, once a week.The AAT did in experimental group,then both groups, there are three post-tests were taken 8th、12th and 16th weeks.
  This scale was adopted in this study to assess the participants' cognitive functions.

SECONDARY OUTCOMES:
The Geriatric Depression Scale (GDS-15) | The experimental and control groups were subjected to a pre-test after they were recruited. There are 12 times AAT, once a week.The AAT did in experimental group,then both groups, there are three post-tests were taken 8th、12th and 16th weeks.
  The two scales were adopted in this study to assess the participants' depressive and the participants' emotion state
The Barthel Index | The experimental and control groups were subjected to a pre-test after they were recruited. There are 12 times AAT, once a week.The AAT did in experimental group,then both groups, there are three post-tests were taken 8th、12th and 16th weeks.
  This index was adopted in this study to assess the participants' physical mobility and function.
The Brief Symptom Rating Scale(BSRS-5) | The experimental and control groups were subjected to a pre-test after they were recruited. There are 12 times AAT, once a week.The AAT did in experimental group,then both groups, there are three post-tests were taken 8th、12th and 16th weeks.
  The participants' feeling healthy

CONTACTS AND LOCATIONS:
Overall Officials: Su-Jen Wang, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
We don't have a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Lai NM, Chang SMW, Ng SS, Tan SL, Chaiyakunapruk N, Stanaway F. Animal-assisted therapy for dementia. Cochrane Database Syst Rev. 2019 Nov 25;2019(11):CD013243. doi: 10.1002/14651858.CD013243.pub2. PMID 31763689
- [Result] Chen H, Wang Y, Zhang M, Wang N, Li Y, Liu Y. Effects of animal-assisted therapy on patients with dementia: A systematic review and meta-analysis of randomized controlled trials. Psychiatry Res. 2022 Aug;314:114619. doi: 10.1016/j.psychres.2022.114619. Epub 2022 May 10. PMID 35623240
- See also: Animal-Assisted Therapy used in psychiatric symptoms and dementia patinets. — https://doi.org/10.6142/VGHN.202012_37(4).0003
- See also: Functional Outcomes in a Randomized Controlled Trial of Animal-Assisted Therapy on Middle-Aged and Older Adults with Schizophrenia. — https://doi.org/10.3389/fpsyt.2021.713623
- See also: Animal-assisted therapy for dementia — https://pubmed.ncbi.nlm.nih.gov/31763689/
- See also: Effects of animal-assisted therapy on patients with dementia: A systematic review and meta-analysis of randomized controlled trials — https://pubmed.ncbi.nlm.nih.gov/35623240/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT06722144/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT06722144/ICF_001.pdf